CLINICAL TRIAL: NCT02254226
Title: A Randomised, Open-label Four-way Crossover Study to Evaluate Pharmacokinetics of Salmeterol (Serevent®) After Inhalation of a 25 μg and 50 μg Single Dose (Metered Dose Inhaler) and a 50 μg and 100 μg Single Dose (Diskus®) in Healthy Male Volunteers
Brief Title: Pharmacokinetics of Salmeterol (Serevent®) After Inhalation With Metered Dose Inhaler (MDI) and Diskus® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1184.8
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (4):
- Salmeterol MDI low (Experimental)
  Interventions: Drug: Salmeterol MDI low
- Salmeterol MDI high (Active Comparator)
  Interventions: Drug: Salmeterol MDI high
- Salmeterol Diskus low (Experimental)
  Interventions: Drug: Salmeterol Diskus low
- Salmeterol Diskus high (Experimental)
  Interventions: Drug: Salmeterol Diskus high

INTERVENTIONS:
Drug: Salmeterol Diskus low
  Arms: Salmeterol Diskus low
Drug: Salmeterol Diskus high
  Arms: Salmeterol Diskus high
Drug: Salmeterol MDI low
  Arms: Salmeterol MDI low
Drug: Salmeterol MDI high
  Arms: Salmeterol MDI high

SUMMARY:
1. To compare the systemic drug exposure of 100 μg Serevent ® Diskus ® with that of 50 μg Serevent ® MDI with sufficient precision so that in combination with a second trial it can be demonstrated that the systemic drug exposure of a new formulation of salmeterol xinafoate is not superior to that of Serevent ® MDI
2. To test a system of ordered null hypotheses regarding the exposure of two dose levels of Serevent ® Diskus ® and Serevent ® MDI
3. To get data about the systemic drug exposure of 25 μg Serevent ® MDI and of 50 μg Serevent ® Diskus ®

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG (electrocardiogram) , clinical laboratory tests 1.1 No finding deviating from normal and of clinical relevance 1.2 No evidence of a clinically relevant concomitant disease
2. Age ≥21 and ≤50 years
3. BMI ≥18.5 and <30 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation.

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts.
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
7. Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to administration or during the trial.
8. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial.
9. Participation in another trial with an investigational drug within 2 months prior to administration or during the trial.
10. Smoker (more than 10 cigarettes or three cigars or three pipes per day)
11. Inability to refrain from smoking on trial days
12. Alcohol abuse (more than 60 g/day)
13. Drug abuse
14. Blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
15. Excessive physical activities (within 1 week prior to administration or during the trial)
16. Any laboratory value outside the reference range that is of clinical relevance
17. Inability to comply with dietary regimen of study centre

    Exclusion criterion specific for this study:
18. Asthma or history of pulmonary hyperreactivity
19. Allergy / hypersensitivity to Lactose monohydrate
20. Hyperthyrosis
21. Allergic rhinitis in need of treatment
22. Cardiac arrhythmia
23. Paroxysmal tachycardia (> 100 beats per minute)
24. Aortic stenosis

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2004-11; Primary Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 6 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | Up to 6 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | Up to 6 hours after drug administration
AUCt1-t2 (Area under the concentration time curve of the analyte in plasma over the time interval t1 to t2) | Up to 6 hours after inhalation
tmax (time from dosing to the maximum concentration of the analyte in plasma) | Up to 6 hours after drug administration
λz (terminal rate constant in plasma) | Up to 6 hours after drug administration
t½ (terminal half-life of the analyte in plasma) | Up to 6 hours after drug administration
MRTinh (mean residence time of the analyte in the body after inhalational administration) | Up to 6 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | Up to 6 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | Up to 6 hours after drug administration
Aet1-t2 (amount of analyte that was eliminated in urine from the time interval t1 to t2) | Up to 6 hours after inhalation
fet1-t2 (fraction of administered drug excreted unchanged in urine from time point t1 to t2) | Up to 6 hours after inhalation
CLR,t1-t2 (renal clearance of the analyte in plasma from the time point t1 to t2) | Up to 6 hours after inhalation
Number of participants with abnormal findings in physical examination | Up to 15 days after last drug administration
Number of participants with clinically significant changes in vital signs | Up to 15 days after last drug administration
Number of participants with abnormal findings in ECG | Up to 15 days after last drug administration
Number of participants with abnormal changes in clinical laboratory parameters | Up to 15 days after last drug administration
Number of participants with adverse events | Up to 15 days after last drug administration